CLINICAL TRIAL: NCT01079377
Title: Psychological Symptoms Among Adolescents Enrolled in a Bariatric Surgery Program
Status: Completed | Type: Observational
Sponsor: New York State Psychiatric Institute (Other)
Responsible Party: Principal Investigator, Leora David, Research Scientist, New York State Psychiatric Institute
Other Study IDs: #6035/#7001R
Record Dates: First submitted 2010-03-02; First posted 2010-03-03 (Estimated); Last update posted 2018-08-23 (Actual); Status verified 2018-08

CONDITIONS: Obesity
Keywords: Adolescents; Bariatric Surgery; Psychological Symptoms; Cognitive Behavioral Therapy; Telemedicine; Longitudinal
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Adolescent Surgical Candidates: Adolescents at the Center for Adolescent Bariatric Surgery, Columbia University Medical Center
- Obese Treatment-Seeking Adolescents: Obese Treatment-Seeking Adolescents, Maxcor Program for Overweight Education and Reduction (POWER) Program
- Normal-Weight Adolescents: Normal-Weight Adolescents

SUMMARY:
This study will examine the interaction of psychological factors and serious overweight to determine if particular patterns of psychological symptoms are helpful in predicting outcomes of weight loss surgery.

Patients from the Center of Adolescent Bariatric Surgery (CABS) program at the Morgan Stanley Children's Hospital of New York Presbyterian will be asked to participate in a longitudinal prospective study of psychopathology among severely obese adolescents. Additionally, the psychological symptoms of this group will be compared to other treatment-seeking obese adolescents.

The investigators hypothesize that:

1. Adolescents receiving bariatric surgery will demonstrate significant reductions in body weight, eating pathology, and other symptoms after receiving bariatric surgery.
2. Adolescents enrolled in the bariatric surgery program will report more psychological problems than other treatment-seeking obese adolescents.

DETAILED DESCRIPTION:
With increasing rates of overweight and obesity among children and adolescents in the United States, there is an urgent need for effective weight loss treatments for younger patients. Recently, bariatric surgery has been considered as a treatment for seriously overweight adolescents because of the potential for substantial decreases in weight and subsequent improvements in physical health. This study will examine the interaction of psychological factors and serious overweight to determine if particular patterns of psychological symptoms (psychological phenotypes) are helpful in predicting outcomes of bariatric surgery. Patients from the Center for Adolescent Bariatric Surgery (CABS) program at the Morgan Stanley Children's Hospital of New York Presbyterian will be asked to participate in a longitudinal prospective study of psychopathology among severely obese adolescents. The final aim of this project is to compare psychological symptoms between obese adolescents seeking bariatric surgery, other treatment-seeking obese adolescents, and normal-weight comparison adolescents. We will evaluate the effect of psychiatric symptoms on adherence to postsurgery follow-up appointments and weight loss. This research will be broadly applicable to the study of interactions between psychological factors and compliance with treatment for youth with chronic health conditions.

ELIGIBILITY:
Longitudinal assessments:

Inclusion Criteria:

* enrolled in the Center for Adolescent Bariatric Surgery (CABS) at the Morgan Stanley Children's Hospital of New York Presbyterian
* entered the CABS program between the ages of 12 and 17, between the ages of 12 and 18 when entering the study
* adolescents speak English
* parents speak English or Spanish

Exclusion Criteria:

* DSM-IV Diagnosis of Mild, Moderate, or Severe Mental Retardation (e.g., IQ < 70)

CONTROL GROUP (obese treatment-seeking adolescents)

Inclusion Criteria:

* enrolled in the Maxcor Program for Overweight Education and Reduction (POWER) Program
* Between the ages of 14 and 18
* adolescents speak English
* parents speak English or Spanish

Exclusion Criteria:

* DSM-IV Diagnosis of Mild, Moderate, or Severe Mental Retardation (e.g., IQ < 70)

CONTROL GROUP (normal-weight adolescents)

Inclusion Criteria:

* body mass index between 25th and 85th percentile for sex
* between the ages of 14 and 18
* adolescents speak English
* parents speak English

Exclusion Criteria:

* DSM-IV Diagnosis of Mild, Moderate, or Severe Mental Retardation (e.g., IQ < 70)

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Adolescent Surgical Candidates, Obese Comparison Subjects, Normal-Weight Comparison Subjects
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2010-01; Primary Completion 2017-01 (Actual); Study Completion 2017-01-05 (Actual)

PRIMARY OUTCOMES:
Psychological Symptoms | 8 assessment points: (1) baseline pre-surgery, (2) 2 weeks pre-surgery, (3) 3 months post-surgery, (4) 6 months post-surgery, (5) 9 months post-surgery, (6) 12 months post-surgery, (7) 18 months post-surgery, (8) 24 months post-surgery
  The measures of psychological symptoms at each time point will include:
  1. Eating and Activity Measures
  2. Depressive Symptom Measures
  3. Impulsivity Measures
  4. Measures of other relevant factors, including body mass index, family functioning, and quality of life.

SECONDARY OUTCOMES:
Treatment Compliance | 8 assessment points: (1) Baseline pre-surgery, (2) 2 weeks pre-surgery, (3) 3 months post-surgery, (4) 6 months post-surgery, (5) 9 months post-surgery, (6) 12 months post-surgery, (7) 18 months post-surgery, (8) 12 months post-surgery
  Clinician rated measures of compliance and adherence to treatment recommendations.

CONTACTS AND LOCATIONS:
Overall Officials: Robyn Sysko, Ph.D., Principal Investigator — New York State Psychiatric Institute
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States